CLINICAL TRIAL: NCT00720772
Title: The Treatment Effect of Intravenous Sodium Thiosulfate on Coronary Calcification in Patients on Hemodialysis
Brief Title: Intravenous Sodium Thiosulfate on Coronary Calcification in Patients on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Sinee Disthabanchong, M.D., Ramathibodi Hospital. Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 02-51-31
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Calcification; Vascular Calcification
Keywords: coronary calcification; vascular calcification; sodium thiosulfate
MeSH Terms: conditions — Vascular Calcification | interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: 25% intravenous (IV) sodium thiosulfate
- B (No Intervention)

INTERVENTIONS:
Drug: 25% intravenous (IV) sodium thiosulfate — 50 ml IV drip twice/week post hemodialysis
  Arms: A

SUMMARY:
The present study will examine the treatment effect of sodium thiosulfate on coronary calcification in patients on hemodialysis.

DETAILED DESCRIPTION:
Coronary calcification (CAC) is prevalent among patients with end-stage renal disease (ESRD). High serum phosphate, the intake of calcium containing phosphate binder as well as dialysis vintage have been shown to be associated with the increasing prevalence of CAC. High CAC score examined by electron-beam CT scan or multi-slice CT scan associates with an increased cardiovascular mortality in ESRD. In series of case reports, intravenous sodium thiosulfate (STS) reduced the calcium burden in calcific uremic arteriopathy and soft tissue calcification. This was believed to be due to the calcium chelation effect of STS.

ELIGIBILITY:
Inclusion Criteria:

* CAC score > 300
* Life expectancy > 6 months
* Dialysis vintage > 6 months

Exclusion Criteria:

* Non-compliance to hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
CAC score | 6 months

SECONDARY OUTCOMES:
Bone mineral density, calcium removal | 6 months, 1 and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sinee Disthabanchong, M.D., Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Phayathai, Bangkok, Thailand

REFERENCES:
- [Background] Goodman WG, Goldin J, Kuizon BD, Yoon C, Gales B, Sider D, Wang Y, Chung J, Emerick A, Greaser L, Elashoff RM, Salusky IB. Coronary-artery calcification in young adults with end-stage renal disease who are undergoing dialysis. N Engl J Med. 2000 May 18;342(20):1478-83. doi: 10.1056/NEJM200005183422003. PMID 10816185
- [Background] London GM, Guerin AP, Marchais SJ, Metivier F, Pannier B, Adda H. Arterial media calcification in end-stage renal disease: impact on all-cause and cardiovascular mortality. Nephrol Dial Transplant. 2003 Sep;18(9):1731-40. doi: 10.1093/ndt/gfg414. PMID 12937218
- [Background] Matsuoka M, Iseki K, Tamashiro M, Fujimoto N, Higa N, Touma T, Takishita S. Impact of high coronary artery calcification score (CACS) on survival in patients on chronic hemodialysis. Clin Exp Nephrol. 2004 Mar;8(1):54-8. doi: 10.1007/s10157-003-0260-0. PMID 15067517
- [Background] Cicone JS, Petronis JB, Embert CD, Spector DA. Successful treatment of calciphylaxis with intravenous sodium thiosulfate. Am J Kidney Dis. 2004 Jun;43(6):1104-8. doi: 10.1053/j.ajkd.2004.03.018. PMID 15168392